CLINICAL TRIAL: NCT00001186
Title: Psychological Benefits of a Normalized Camping Experience for Children With Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 830022; 83-C-0022; NCT00018915 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-05-23

CONDITIONS: Pediatric Cancer
Keywords: Psychosocial; Self Esteem; Oncology; Well-Being; Pediatrics; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Children 7-17 years of age who are currently being treated for cancer or are up to 5 years post therapy.
- Cohort 2: Young adults with cancer (YACers) 18-25 years of age acting as counselors at Camp Fantastic and are enrolled in another NIH protocol.

SUMMARY:
Background:

* Cancer has an enormous impact on the psychological and social well-being of the family unit. The life-threatening connotations of cancer single out the ill child from his peer/family group as one who is different, and often unable to maintain a normal lifestyle. Physical sequelae of cancer and its treatment accentuate the differences between these children and their normal peers/siblings.
* It is important that children with cancer be prepared to function outside of protected situations and begin to develop skills of separation and independence. For healthy children, some of these latter skills are acquired by a camping experience. Such an experience for the patient with cancer is frequently precluded by their dependence on medical facilities and the physical limitations of their activities.
* The goal of this study will be to assess the short and long term benefits of the "normalized" camping experience, provided in conjunction with Special Love, Inc., on the patients and staff. In particular, we will seek to determine whether such a comprehensive experience is capable of influencing the attitudes and life experiences of patients and staff in a positive manner.

Objectives:

-To evaluate the impact of an enriched normalized camping experience on the quality of life of the pediatric cancer patient. In particular, attempts will be made to measure the manner in which this experience influences the child's sense of well-being and self-esteem as well as his or her relationship with parents, family, and peers.

Eligibility:

* Children 7-17 years of age who are currently being treated for cancer or are up to 3 years post therapy OR Young adults with cancer (YACers) 18-25 years of age who are acting as counselors at Camp Fantastic
* All children/young adults will be selected for camp after careful screening by a multidisciplinary committee consisting of medical and program directors.
* At the discretion of the multidisciplinary committee consisting of medical and program directors, special exceptions may be made for children with extenuating circumstances.

Design:

* Assessment of benefit may include interviews with children and families before, during and following camp. Observational data on the child's performance at camp will be noted.
* Medical and nursing personnel will consist of staff from the Pediatric Branch at the NCI, other units within the NIH, and participating institutions.
* Special Love members, the Program Director at the 4-H Center camp (site of the camp) and Pediatric Branch staff at the NCI will coordinate the camp program, taking into account the medical needs of each camper.
* Every attempt will be made to provide a full agenda of age appropriate activities for the patients.
* The length of the camping experience for children with cancer will be for 7 days beginning on a Sunday and extending through the following Saturday morning. Patients will be transported to the camp from the NIH Clinical Center and the Virginia hospitals by bus.

DETAILED DESCRIPTION:
Background:

* Cancer has an enormous impact on the psychological and social well-being of the family unit. The life-threatening connotations of cancer single out the ill child from his peer/family group as one who is different, and often unable to maintain a normal lifestyle. Physical sequelae of cancer and its treatment accentuate the differences between these children and their normal peers/siblings.
* It is important that children with cancer be prepared to function outside of protected situations and begin to develop skills of separation and independence. For healthy children, some of these latter skills are acquired by a camping experience. Such an experience for the patient with cancer is frequently precluded by their dependence on medical facilities and the physical limitations of their activities.
* The goal of this study will be to assess the short and long term benefits of the "normalized" camping experience, provided in conjunction with Special Love, Inc., on the patients and staff. In particular, we will seek to determine whether such a comprehensive experience is capable of influencing the attitudes and life experiences of patients and staff in a positive manner.

Objectives:

-To evaluate the impact of an enriched normalized camping experience on the quality of life of the pediatric cancer patient. In particular, attempts will be made to measure the manner in which this experience influences the child's sense of well-being and self-esteem as well as his or her relationship with parents, family, and peers.

Eligibility:

* Children 7-17 years of age who are currently being treated for cancer or are up to 5 years post therapy OR Young adults with cancer (YACers) 18-25 years of age who are acting as counselors at Camp Fantastic and are enrolled in another NIH protocol.
* All children/young adults will be selected for camp after careful screening by a multidisciplinary committee consisting of medical and program directors.
* At the discretion of the multidisciplinary committee consisting of medical and program directors, special exceptions may be made for children with extenuating circumstances.

Design:

* Assessment of benefit may include interviews with children and families before, during and following camp. Observational data on the child's performance at camp will be collected.
* Medical and nursing personnel will consist of staff from the Pediatric Oncology Branch at the NCI, other units within the NIH, and participating institutions.
* Special Love members, the Program Director at the 4-H Center camp (site of the camp) and Pediatric Oncology Branch staff at the NCI will coordinate the camp program, taking into account the medical needs of each camper.
* Every attempt will be made to provide a full agenda of age appropriate activities for the patients.
* The length of the camping experience for children with cancer will be for 7 days beginning on a Sunday and extending through the following Saturday morning. Patients will be transported to the camp from the NIH Clinical Center and the Virginia hospitals by bus.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Children 7-17 years of age who are currently being treated for cancer or are up to 5 years post therapy.

OR

Young adults with cancer (YACers) 18-25 years of age who are acting as counselors at Camp Fantastic.

* Children/young adults will be selected for camp after careful screening by a multidisciplinary committee consisting of medical and program directors. While the state of the child s health will certainly be considered there will be no exclusions for:
* Patients who are receiving intramuscular, intrathecal, oral or intravenous medications or blood products.
* Patients who have had amputations or have other physical defects.
* Patients who become febrile and neutropenic at the onset or during the week of camp will stay at camp on antibiotic therapy providing their condition remains stable.
* At the discretion of the multidisciplinary committee consisting of medical and program directors, special exceptions may be made for patients with extenuating circumstances.
* All children will be officially enrolled and will have an NIH Clinical Center Patient Care Number. The enrollment of a child, signing of protocol consent, and completion of admission paperwork is done in person but under extenuating circumstances it may be done over the phone after the paperwork has been mailed to the parent/guardian. Extenuating circumstances would include a last minute application to camp after the trip for camp screenings in Norfolk or Richmond has been completed.

EXCLUSION CRITERIA:

-Children with a medical diagnosis other than cancer or their related disorders.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 7-17 years of age who are currently being treated for cancer or are up to 5 years post therapy, OR, Young Adults with Cancer (YACers) 18-25 years of age who are acting as counselors at Camp Fantastic and are enrolled in another NIH protocol.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1983-02-15 (Actual)

PRIMARY OUTCOMES:
Increase in self esteem | Ongoing
  Psychological benefit

SECONDARY OUTCOMES:
Improvement in quality of interactions | ongoing
  Psychological benefit

CONTACTS AND LOCATIONS:
Overall Officials: John F Shern, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
BTRIS: All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: BTRIS: Clinical data available during the study and indefinitely.
Access Criteria: BTRIS: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Weissman MM, Orvaschel H, Padian N. Children's symptom and social functioning self-report scales. Comparison of mothers' and children's reports. J Nerv Ment Dis. 1980 Dec;168(12):736-40. doi: 10.1097/00005053-198012000-00005. PMID 7452212
- [Background] Reinhard SC, Given B, Petlick NH, Bemis A. Supporting Family Caregivers in Providing Care. In: Hughes RG, editor. Patient Safety and Quality: An Evidence-Based Handbook for Nurses. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Apr. Chapter 14. Available from http://www.ncbi.nlm.nih.gov/books/NBK2665/ PMID 21328765
- [Background] Achenbach TM, Edelbrock CS. The Child Behavior Profile: II. Boys aged 12-16 and girls aged 6-11 and 12-16. J Consult Clin Psychol. 1979 Apr;47(2):223-33. doi: 10.1037//0022-006x.47.2.223. No abstract available. PMID 469068
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1983-C-0022.html